CLINICAL TRIAL: NCT01599377
Title: Phase 1, Open-Label, Randomized, Single-Dose, Cross-Over, Bioequivalence Study Comparing Tablets (5 And 10 Mg) And Capsules (5 And 10 Mg) Of Tofacitinib Under Fasted Conditions In Healthy Volunteers
Brief Title: Tofacitinib Bioequivalence Study Comparing Tablets And Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A3921141
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: tofacitinib 10 mg
- Cohort 2 (Experimental)
  Interventions: Drug: tofacitinib 5 mg

INTERVENTIONS:
Drug: tofacitinib 10 mg — Cohort 1 will consist of 2 periods and 2 sequences. Subjects will be randomized to one of the 2 sequences. In sequence 1, subjects will receive a 10 mg tofacitnib tablet under fasting conditions in period 1, followed by a 10 mg tofacitinib capsule in fasting conditions in period 2. In sequence 2, the treatments will be reversed for period 1 and 2.
  Arms: Cohort 1
Drug: tofacitinib 5 mg — Cohort 2 will consist of 2 periods and 2 sequences. A total of 24 healthy subjects will be enrolled for this cohort. Subjects will be randomized to one of the 2 sequences. In sequence 1, subjects will receive a 5 mg tablet under fasting conditions in period 1, followed by a 5 mg capsule in fasting conditions in period 2. In sequence 2, the treatments will be reversed for period 1 and 2.
  Arms: Cohort 2

SUMMARY:
The overall aim of the study is to establish bioequivalence between commercial tofacitinib tablet formulations with the tofacitinib capsule formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non-childbearing potential) subjects between the ages of 21 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including oral temperature, BP and PR measurement, 12 Lead ECG and clinical laboratory tests.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf ) | 24 hours
Maximum plasma concentration (Cmax) | 24 hours

SECONDARY OUTCOMES:
Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (AUClast) | 24 hours
Time for Cmax (Tmax) | 24 hours
Terminal elimination half-life (t½) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921141&StudyName=Tofacitinib%20Bioequivalence%20Study%20Comparing%20Tablets%20And%20Capsules